CLINICAL TRIAL: NCT06251960
Title: Comparison of Autogenous Completely Demineralized Dentin Graft Versus Partially Demineralized Dentin Graft Used in Preservation of Post-Extraction Sites Associated With Delayed Implant Placement
Brief Title: Demineralized Dentin Graft in Preservation of Post-Extraction Sites Associated With Delayed Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A01012023OS
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-01

CONDITIONS: Socket Preservation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- socket preservation with completely demineralized dentin graft. (Experimental)
  Interventions: Procedure: socket preservation with completely demineralized dentin graft
- socket preservation with partially demineralized dentin graft. (Experimental)
  Interventions: Procedure: socket preservation with partially demineralized dentin graft

INTERVENTIONS:
Procedure: socket preservation with completely demineralized dentin graft — socket preservation with completely demineralized dentin graft followed by delayed implant placement after 4 months
  Arms: socket preservation with completely demineralized dentin graft.
Procedure: socket preservation with partially demineralized dentin graft — socket preservation with completely demineralized dentin graft followed by delayed implant placement after 4 months
  Arms: socket preservation with partially demineralized dentin graft.

SUMMARY:
Thirty patients will be selected from outpatient clinic of the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University seeking for extraction of non-restorable mandibular posterior teeth For the 1st group: the socket will be grafted with completely demineralized dentin graft after 3 days of extraction, followed by delayed implant placement after 4 months.

For the 2nd group: the socket will be grafted with partially demineralized dentin graft in in the same day of extraction, followed by delayed implant placement after 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient medically free from systemic diseases.
* Patient with good oral hygiene.
* Age above 18 years.
* Presence of non-restorable mandibular premolar tooth due to caries, root resorption, roots fracture, etc.
* No acute infection is present.
* No history of bruxism.
* Patients prepared to comply with the follow-up and maintenance program.

Exclusion Criteria:

* Patients with systemic diseases that interfere with dental implant insertion.
* Pregnancy.
* Immunocompromised patients.
* Existence of non-treated generalized progressive periodontitis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Histomorphometric evaluation: | 4 monhs
  After 4 months of socket preservation and just before implant placement, a trephine bur will be used to collect a core of bone from the preserved socket. Bone will be examined histologically to evaluate the quality and quantity of the formed bone.
  Briefly, the specimens were fixed with 4% paraformaldehyde in 0.1M PBS (pH 7.4) and decalcified in 0.5M EDTA (pH 7.8). After decalcification, each specimen will be processed and embedded in paraffin, and transverse serial sections of 5 μm thickness will be prepared. The sections will be stained with hematoxylin and eosin (H&E), Masson's Trichrome (MT) (Cat # HT15, Sigma Aldrich) and immunohistochemical staining with osteocalcin antibody polyclonal osteocalcin (OCN);diagnostic biosystems), histological examination will be carried out using an Olympus BX-51 optical microscope (Olympus Co., Tokyo, Japan).
Histomorphometric analysis | 4 months
  Microscopic images of the surgical sites will be taken by randomly selecting four areas of the center portion of the defect at 100× magnification. Then, using 16 images of each group, the ratio of newly formed bone to the entire defect area in the slide images will be calculated in trichrome and osteocalcin-stained images using the Intel® Core I7® based computer using VideoTest Morphology® software (Russia) with a specific built-in routine for % area, measurement.
Bone density: | 12 months
  Bone density will be evaluated using Cone Beam Computed Tomography (CBCT) that will be made immediately after socket preservation, at 4 months after preservation (just before implant placement), and after 12 months from implant loading.

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Elsheikh, Al Mansurah, Egypt